CLINICAL TRIAL: NCT06048705
Title: Assessment of Safety and Recommended Phase 2 Dose of Autologous T Cells Engineered With an Affinity-enhanced TCR Targeting NYESO1 and LAGE1a, and Co-expressing CD8α (GSK3901961) in Participants With NYESO1 and/or LAGE1a Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma / Myxoid/Round Cell Liposarcoma; or NYESO1 and/or LAGE1a Positive Previously Treated Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of GSK3901961 In Previously Treated Advanced (Metastatic OR Unresectable) Synovial Sarcoma/ Myxoid/Round Cell Liposarcoma, and Previously Treated Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in GSK's R&D priorities.
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209012 Substudy 1
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: Adoptive T cell therapy; Advanced synovial sarcoma; Advanced Myxoid/Round Cell Liposarcoma; Advanced tumors; GSK3901961; T cell receptor; Leukapheresis; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Liposarcoma, Myxoid; Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK3901961 (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive high dose of GSK3901961 after completing lymphodepleting chemotherapy. The first study participant receiving GSK3901961 will receive the total assigned dose as 2 separate infusions 7 days apart, in aliquots of 30% (first infusion) and 70% (second infusion) of the total target dose, respectively. Based on the dose limiting toxicities reported in the first participant, then all subsequent participants treated with GSK3901961 will receive the full dose as a single, i.e., one-time, infusion.
  Interventions: Drug: GSK3901961; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: GSK3901961 — GSK3901961 was administered.
Drug: Cyclophosphamide — Cyclophosphamide was administered as lymphodepleting chemotherapy.
Drug: Fludarabine — Fludarabine was administered as lymphodepleting chemotherapy.

SUMMARY:
The primary purpose of this sub study is to assess the safety, tolerability and determine recommended Phase 2 dose (RP2D) of GSK3901961 in HLA A*02:01, HLA-A*02:05 and/or HLA A*02:06 positive participants with New York esophageal squamous cell carcinoma (NY ESO 1) and/or Cancer testis antigen 2 (LAGE 1a) positive previously treated metastatic Non-Small Cell Lung Cancer (NSCLC) and previously treated, advanced (metastatic or unresectable) Synovial Sarcoma/ Myxoid/Round Cell Liposarcoma SS/MRCLS.

DETAILED DESCRIPTION:
This study is a substudy of the Master record - (209012) NCT04526509.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be >=18 years of age and weighs ≥40 kg on the day of signing informed consent
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles
* Participant's tumor must have tested positive for NY-ESO-1 and/or LAGE-1a expression by a GSK designated laboratory
* Performance status: Eastern Cooperative Oncology Group of 0-1
* Participant must have adequate organ function and blood cell counts 7 days prior to leukapheresis
* Participant must have measurable disease according to RECIST v1.1.
* Participant has advanced (metastatic or unresectable) SS or MRCLS confirmed by local histopathology with evidence of disease-specific translocation
* Participant has completed at least one standard of care (SOC) treatment including anthracycline containing regimen unless intolerant to or ineligible to receive the therapy.
* Participants who are not candidates to receive anthracycline should have received ifosfamide unless also intolerant to or ineligible to receive ifosfamide. Participants who received neoadjuvant/adjuvant anthracycline or ifosfamide based therapy and progressed will be eligible
* Participant has histologically or cytologically confirmed Stage IV NSCLC
* Participant has been previously treated with SOC for Stage IV NSCLC

Exclusion Criteria:

* Central nervous system (CNS) metastases, with certain exceptions for CNS metastases in NSCLC as specified in the protocol
* Any other prior malignancy that is not in complete remission
* Clinically significant systemic illness
* Prior or active demyelinating disease
* History of chronic or recurrent (within the last year prior to leukapheresis) severe autoimmune or immune mediated disease requiring steroids or other immunosuppressive treatments
* Previous treatment with genetically engineered NY-ESO-1-specific T cells, NY-ESO-1 vaccine or NY-ESO-1 targeting antibody
* Prior gene therapy using an integrating vector
* Previous allogeneic hematopoietic stem cell transplant within the last 5 years or solid organ transplant
* Washout periods for prior radiotherapy and systemic chemotherapy must be followed
* Major surgery within 4 weeks prior to lymphodepletion
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaptimmune Patient Enquiries, Principal Investigator — Adaptimmune
Locations (20):
- United States (11):
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: http://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a sub study of the master protocol (NCT04526509). The study was terminated due to a change in GSK's R&D priorities.
Groups:
- GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 1 × 10^9 - 8 × 10^9 cells of GSK3901961 as an intravenous (IV) infusion in two aliquots (approximately 30% on Day 1 and approximately 70% on Day 8) for sentinel participant after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 0.1 × 10^9 - 0.8 × 10^9 cells of GSK3901961 as an intravenous (IV) infusion on Day 1 after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- No Treatment: No Treatment arm consisted of participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy and T cell infusion.
Period: Overall Study
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment
Started | 1 | 4 | 2
Transferred to Long-term Follow-up Study | 0 | 2 | 0
Death Post Lymphodepletion | 0 | 2 | 0
Completed (Participants who were transferred to the long-term follow-up protocol or have died are considered to have completed.) | 0 | 4 (2 participants transferred to long-term follow-up study 208750 (NCT03391778) and 2 participants died post lymphodepletion.) | 0
Not Completed | 1 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Did not meet Inclusion/Exclusion Criteria | 0 | 0 | 1
Not completed — Death prior to lymphodepletion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment | Total
Number analyzed (Participants) | 1 | 4 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 | 51.5 (17.79) | 43.0 (0.00) | 45.6 (15.53)
Age, Customized [Count of Participants; unit: Participants]
  Age, customized: 19-64 | 1 | 3 | 2 | 6
  Age, customized: >=65 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 0 | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 4 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 4 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Australia | 0 | 1 | 0 | 1
  Germany | 0 | 2 | 1 | 3
  Sweden | 0 | 1 | 0 | 1
  United States | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT events were graded according to NCI-CTCAE v5.0. DLTs were defined as Grade (Gr) 4 (life-threatening and death) related to GSK3901961 2) Gr 3 (Severe or medically significant) at least possibly related to GSK3901961 and do not resolve to Gr <=1 (or Baseline) within 7 days from the onset of the event 3) Gr >=3 non-infectious pneumonitis not responding to oxygen supplementation and systemic steroid treatment 4) Any Gr 3 cytokine release syndrome (CRS) at least possibly related to GSK3901961 that does not improve to Gr <2 (moderate) toxicity within 7 days with or without dexamethasone 5) Any Gr 4 CRS at least possibly related to study product that does not improve to Gr <=2 (or Baseline) within 7 days 6) Any Gr 3 or greater neurotoxicity that does not resolve to Gr <=2 within 72 hours 7) Any Gr >=3 organ toxicity (exclusive of CRS toxicity) involving major organ systems that persists for >72 hours and occurs within 28 days of infusion.
Time Frame: Up to 28 days
Population: DLT Evaluable included participants in the mITT population (all ITT participants (All participants who started leukapheresis procedure) who received any dose of New York esophageal antigen-1 [NY ESO 1] specific T cells) who are part of the dose confirmation phase that either had a DLT or have completed the DLT assessment period of 28 days since last T cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
Participants | 1 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs Based on Maximum Severity
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE is defined as any untoward medical occurrence that, at any dose can result in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth or is medically significant or requires intervention to prevent one or the outcomes listed above. AEs and SAEs were graded according to NCI-CTCAE v5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE. AEs which start or worsen on or after T-cell infusion are classified as treatment emergent. SAEs are subset of AEs. Results for maximum severity grades has been presented.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population included all ITT participants (All participants who started leukapheresis procedure) who received any dose of NY ESO 1 specific T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
Participants
  AEs, Grade 1 | 0 | 0
  AEs, Grade 2 | 0 | 0
  AEs, Grade 3 | 0 | 0
  AEs, Grade 4 | 1 | 3
  AEs, Grade 5 | 0 | 1
  SAEs, Grade 1 | 0 | 1
  SAEs, Grade 2 | 0 | 0
  SAEs, Grade 3 | 1 | 0
  SAEs, Grade 4 | 0 | 0
  SAEs, Grade 5 | 0 | 1

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events of Special Interest (AESI)
Description: An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included events of Cytokine Release Syndrome (CRS), Haematopoietic cytopenias (including pancytopenia and aplastic anaemia), Graft versus Host Disease (GvHD), Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS), Guillain-Barre Syndrome (GBS), Pneumonitis and treatment-related inflammatory response at tumor site(s) and Neutropenia Grade 4 lasting more than or equal to 28 days. AEs which start or worsen on or after T-cell infusion are classified as treatment emergent.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
Participants
  Participants with any AESI | 1 | 4
  Cytokine Release Syndrome (CRS) | 1 | 3
  Graft versus host disease | 1 | 0
  Haematopoietic cytopenias (including pancytopenia and aplastic anaemia) | 1 | 4
  Immune Effector-Cell Associated Neurotoxicity Syndrome | 0 | 1

4. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator According to RECIST v1.1
Description: Overall response rate (ORR) defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1 relative to the total number of participants in the analysis population. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response (CR) was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
percentage of participants | 100 [2.5 to 100] | 50 [6.8 to 93.2]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the interval of time (in months) from first documented evidence of the confirmed response (PR or CR) as assessed by local investigators to the date of disease progression per RECIST v1.1 or death due to any cause, among participants with a confirmed response of PR or CR. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population. Only responders (CR or PR) by investigator assessment were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 2
Months | 1.22 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the duration of response for this single participant who was censored at their last tumor assessment prior to study withdrawal. | 2.96 [2.8 to 3.1]

6. Secondary Outcome: Maximum Transgene Expansion (Cmax) of GSK3901961
Description: Cmax was defined as peak cell expansion during the interventional phase. Blood samples were collected to measure Cmax.
Time Frame: Up to 21 days
Population: Pharmacokinetic population included participants from the mITT population for whom at least one persistence sample was obtained, analysed, and was measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
Copies per microgram genomic DNA | 121973 (NA) — Geometric coefficient of variation is not applicable as only a single participant was analyzed. Geometric mean value presented here is the actual Cmax. | 29058.02 (401.296)

7. Secondary Outcome: Time to Cmax (Tmax) of GSK3901961
Description: Tmax was defined as time to peak cell expansion during the interventional phase. Blood samples were collected to measure Tmax.
Time Frame: Up to 21 days
Population: Pharmacokinetic population included participants from the mITT population for whom at least one persistence sample was obtained, analyzed, and was measurable.
Measure: Median (Full Range); unit: days
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
days | 21 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual Tmax for this single participant. | 7.5 [1 to 20]

8. Secondary Outcome: Area Under the Time Curve From Zero to Time 28 Days AUC(0-28)
Description: Area under the cell expansion-time curve from first T-cell infusion to Day 28. Blood samples were collected to measure AUC (0-28 days).
Time Frame: Up to 28 days
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies per microgram genomic DNA
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 4
Days*copies per microgram genomic DNA | 2267635.372 (NA) — Geometric coefficient of variation is not applicable as only a single participant was analyzed. Geometric mean value presented here is the actual AUC(0-28). | 374639.00 (371.441)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 21 months.
Description: All-cause mortality, SAEs and non-SAEs were reported for intent-to-treat (ITT) population that included all participants who started leukapheresis procedure.
Arm/Group | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/4 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/4 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells (N=1) | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells (N=4) | No Treatment (N=2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells (N=1) | GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells (N=4) | No Treatment (N=2)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (4) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Interleukin level increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT06048705/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT06048705/SAP_001.pdf